CLINICAL TRIAL: NCT06733870
Title: Peri-implant Soft Tissue and Bone Evaluation of One Abutment One Time Concept Following Fully Computer Guided Immediate Implants
Brief Title: Peri-implant Soft Tissue and Bone Evaluation in Fully Computer Guided Immediate Implants
Acronym: randomised
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nouran Abd El Nasser, Assistant lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: FDASU.REC ID 032124
Record Dates: First submitted 2024-12-01; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Soft Tissue Healing
Keywords: One abutment one time; Full digital workflow; Immediate implant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- immediate load with provisional restoration (Other): immediate load with PMMA crown on Ti base
  Interventions: Procedure: guided immediate implant surgery
- immediate load with one abutment one time concept (Other): immediate ;load with customized final abutment and PMMA crown
  Interventions: Procedure: guided immediate implant surgery

INTERVENTIONS:
Procedure: guided immediate implant surgery — fully guided immediate implant placement and loading

SUMMARY:
Prospective evaluation of perimplant soft tissue and bone response to one abutment one-time concept versus provisional abutment in fully guided single immediate implant placement.

DETAILED DESCRIPTION:
Patient selection:

The study will be conducted on total of 16 patients recruited from the outpatient clinic of Oral Medicine, Periodontology, Oral Diagnosis and Radiology department, Faculty of Dentistry, Ain-Shams University. Sixteen consecutive healthy male/female patients with single non restorable remaining maxillary root from the right second premolar to the left second premolar will be added to the study.

Sample size analysis :

A sample size of 14 (7 in each group) will be sufficient to detect an effect size of approximately 1.75, with a power (1-β error) of 0.8 (80%) using a two-sided hypothesis test, with a significance level (α error) 0.05 for data. G power program version 3.1.9.2 was used for sample size calculation.This was increased to 8 patients in each group to make up for lost follow up cases The procedure will be explained to all patients and an informed consent will be signed before their inclusion in the study.

These patients will be divided randomly into 2 groups:

Group I: will include 8 patients who will undergo guided immediate implant placement and immediate provisionalization with preplanned PMMA provisional restoration on Ti-Base Group II: will include 8 patients who will undergo guided immediate implant placement and immediate loading by using a final CAD/CAM customized abutment and a cemented CAD/CAM fabricated PMMA provisional restoration.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged at least 18 years.
* Patients free from any systemic disease as evidenced by health questionnaire - - Single tooth failure of a maxillary anterior region (incisors, canines, and premolars) with neighbouring teeth present and healthy periodontal conditions.
* Intact socket walls evident on cone beam computed tomography and confirmed on the day of extraction.
* Natural teeth present adjacent to the tooth being replaced in addition to a natural counterpart tooth present for esthetics criteria evaluation.
* Adequate bone apical to the tooth to be replaced with a minimum primary stability of 30 Ncm.
* Thick gingival biotype.

Exclusion Criteria:

* Presence of active infection around the failing tooth or adjacent teeth.
* Presence of active periodontal disease and gingival recession in the esthetic area.
* Systemic diseases , pregnancy and smoking.
* Recent orthodontic treatment.
* Bruxism and parafunctional habits .
* Labial plate dehiscence, fenestration, or loss after tooth extraction
* Inability to achieve primary stability after implant placement
* Vulnerable groups: prisoners, mentally retarded, etc

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2024-02-11 (Actual); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
peri-implant soft tissue volumetric change | 4 months
  * intraoral scanner is used to obtain before and after 3D scans
  * 3D scans are superimposed on a software and the difference in volume can be measured and detected by a color map

SECONDARY OUTCOMES:
Esthetic evaluation | 4 months
  * Esthetic evaluation will be done by calculating the pink esthetic score (PES)
  * standardized photographs are assesed to measure the changes in PES

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Bissar, Associate professor, Study Director — Faculty of dentistry- Ain Shams University; Ingy Nouh, lecturer, Study Director — Faculty of dentistry- Ain Shams University; Hala Kamal, Professor, Study Director — Faculty of dentistry- Ain Shams University
Locations (1):
- faculty of Dentistry ASU, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No